CLINICAL TRIAL: NCT03789032
Title: A Phase 1, Fixed Sequence, Open-label Study in Healthy Adult Subjects to Evaluate the Effect of Multiple Doses of Rabeprazole on the Pharmacokinetics of a Single Dose of Vadadustat
Brief Title: Study to Evaluate the Effect of Rabeprazole on the Pharmacokinetics of Vadadustat
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0033
Record Dates: First submitted 2018-12-27; First posted 2018-12-28 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Drug Interaction Potentiation; Pharmacokinetics
Keywords: Vadadustat; Rabeprazole; Pharmacokinetics
MeSH Terms: interventions — vadadustat; Rabeprazole

STUDY DESIGN:
Intervention Model Description: This is a single arm fixed sequence study. Subjects will be administered vadadustat on day 1, rabeprazole on days 2 to 5, and vadadustat and rabeprazole on day 6.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rabeprazole and Vadadustat (Experimental): Subjects will receive vadadustat 300 mg on day 1, rabeprazole 20 mg every 12 hours on days 2 through 5 and vadadustat 300 mg and rabeprazole on day 6
  Interventions: Drug: Vadadustat; Drug: Rabeprazole

INTERVENTIONS:
Drug: Vadadustat — Vadadustat 300 mg
Drug: Rabeprazole — Oral Rabeprazole

SUMMARY:
This is a Phase 1, fixed sequence, open-label study to evaluate the effect of multiple oral doses of rabeprazole on the pharmacokinetics of a single dose of vadadustat 300 mg in healthy male and female subjects.

DETAILED DESCRIPTION:
This is a Phase 1, fixed sequence, open-label study in healthy adult subjects to evaluate the effect of multiple doses of rabeprazole on the pharmacokinetics of a single dose of vadadustat in healthy male and female subjects. Approximately twenty (20) subjects, with at least 30% female subjects, will be enrolled to ensure 18 evaluable subjects. Subjects will be on study for up to 66 days, including a 28-day screening period, 9-day clinic period, and a 30-day follow- up period post last dose. Subjects who are confirmed eligible and receive at least one dose of study drug will be considered enrolled in the study. Blood samples for PK analysis will be collected at pre-defined time points throughout the study up to 48 hours post administration of vadadustat.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male or female between 18 and 55 years of age, inclusive, at time of informed consent
* Body mass index between 18.0 and 30.0 kg/m2, with a minimum body weight of 45 kg for females and 50 kg for males, inclusive.

Exclusion Criteria:

* Current or past clinically significant history of cardiovascular, cerebrovascular, pulmonary, gastrointestinal, hematologic, renal, hepatic, immunologic, metabolic, urologic, neurologic, dermatologic, psychiatric, or other major disease. History of cancer (except treated non-melanoma skin cancer) or history of chemotherapy use within 5 years prior to Screening.
* Positive test results for human immunodeficiency virus (HIV) antibody; Positive test results of hepatitis B surface antigen (HBsAg), or positive hepatitis C virus antibody (HCVab) within 3 months prior to screening , or positive test results for human immunodeficiency virus antibody (HIVab) at Screening
* Taking any prescription medication or over the counter multi-vitamin supplement, or any non-prescription products (including herbal-containing preparations but excluding acetaminophen) within 14 days prior to Day -1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-19 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from 0 to last quantifiable concentration (AUClast) for vadadustat | Up to 10 weeks
Area under plasma concentration-time curve from 0 to infinity (AUCinf) for vadadustat | Up to 10 weeks
Maximum observed plasma concentration (Cmax) for vadadustat | Up to 10 weeks

SECONDARY OUTCOMES:
Time to maximum observed plasma concentration (Tmax) of vadadustat | Up to 10 weeks
Elimination rate constant (Kel) of vadadustat | Up to 10 weeks
Terminal half-life (t½) of vadadustat | Up to 10 weeks
Apparent total body clearance (CL/F) of vadadustat | Up to 10 weeks
Percent of extrapolated area under the curve from time t to infinity (%AUCextrap) of vadadustat | Baseline and end of study
Area under plasma concentration-time curve from 0 to last quantifiable concentration (AUClast) of vadadustat-O-glucuronide | Up to 10 weeks
Area under plasma concentration-time curve from 0 to infinity (AUCinf) of vadadustat-O-glucuronide | Up to 10 weeks
Maximum observed plasma concentration (Cmax) of vadadustat-O-glucuronide | Up to 10 weeks
Reporting of treatment emergent adverse event (TEAE) as reported by study subjects | Up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Akebia Therapeutics, Study Director — Sponsor GmbH
Locations (1):
- inVentiv Health Clinique Inc., Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided